CLINICAL TRIAL: NCT02252705
Title: Mexican Registry of Pulmonary Hypertension
Acronym: REMEHIP
Status: Completed | Type: Observational
Sponsor: Remehip (Other)
Collaborators: Medicaweb, S.A.C.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: REMEHIP
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary arterial hypertension; Mortality; Survival
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Incident patients: Patients with less than three months from diagnosis to start of the Registry or those who have been diagnosed during the recruitment period.
- Prevalent patients: Patients who have been diagnosed with more than three months from diagnosis to start of the Registry.

SUMMARY:
Prospective multicenter registry including incident patients and prevalent patients which pretends to identify clinical characteristics, treatment trends in-hospital and four years follow-up outcome through major adverse cardiovascular events (MACE) in a Mexican population with well characterized Pulmonary Hypertension.

DETAILED DESCRIPTION:
Introduction. Pulmonary hypertension (PH) is a worldwide group of vascular diseases characterized by progressive increase in pulmonary vascular resistance and pulmonary arterial pressure with secondary vascular and right ventricular (RV) remodeling, RV dysfunction, heart failure syndromes and, finally, premature death. In developed countries significant medical advances have occurred in the last two decades including a more systematic assessment and availability of new therapeutic approaches. In addition, current registries had shown new data regarding epidemiology, demography, clinical presentation, treatment and prognosis. However, the evidence coming from developing countries is scarce and more information is necessary to identify current care in such populations. In the other hand, high quality clinical registries may help to understand if the knowledge coming from clinical trials is being properly applied and if their results are reproducible in day-to-day clinical practice. The results of the REMEHIP, a registry with one-year enrollment and four-year follow-up will hopefully broad the investigators knowledge about clinical profile, medical care, therapeutic trends and outcome in a Mexican population with well characterized PH.

Variables to be included. In all patients: a) date of onset of symptoms, b) medical history, c) personal and family history, c) treatment at enrollment, d) physical examination, d) WHO function class, e) six-minute walk distance, f) ECG, g) chest x-ray, h) echocardiogram, i) pulmonary function tests, j) V/Q lung scan and or pulmonary angiography, and/or pulmonary angiotomography k) right heart catheterization, and whenever possible indicated acute vasodilator challenge 11, 12, l) biomarkers: troponin I (TnI), brain natriuretic peptide (BNP), D - dimer (DD), INR, n) current treatment, o) in-hospital and follow - up outcome, p) MACE.

Visit office. Data will be collected in the first outcome and update through each follow-up about expected PH symptoms, functional class (WHO), current treatment, dose, compliance, collateral effects and concomitant medication, weight, blood pressure, heart and respiratory rate, and biomarkers, when possible or feasible; in patients under oral anticoagulation INR will be recorded in each visit.

Visits will be according with the standard health care of each center, but in general they will be made at least one every six months.

Sites. In centers (outcome treatment and tertiary center), investigators with expertise and experience in diagnosis, stratification and treatment of patients with PH will be involved. Centers without expertise, but with facilities to diagnosis, stratification (six-minute walk distance, pulmonary function tests, V/Q lung scan and or pulmonary angiography, right heart catheterization, and biomarkers) will be included too, as long as they adhere to protocol.

Quality Criteria. Following criteria will be used to improve quality data: a) standardized definitions, data and reports; b) tools for fast feedback; c) meetings among principal investigators and steering committee, at least one per year; d) ethics procedures review; e) electronic, simple and accessible data collection; f) rigorous center selection based on investigators expertise and/or facilities resources); g) consecutive patients enrollment to obtain representative sample; h) random centers audit; i) centralized data and statistical analysis; j) report all data and consistent conclusion; and k) transparency of funds for any publication. Furthermore, the quality of this registry will also be measured by the number of publications and presentations in national and international meetings as has previously been done.

Data collection. Electronic database will have 178 variables including among others, data of onset symptoms, medical history, personal and family history, physical examination, six - minute walk distance, treatment, ECG, chest x-ray, echocardiogram, pulmonary function tests, V/Q lung scan, pulmonary angiography, right heart catheterization, acute vasodilator challenge, biomarkers and (in the follow - up) MACE.

Statistics. Differences between continuous variables with normal distribution will be examined by Student's t test. The test of Wilcoxon rank sum will be used when continuous variables have failed in normality tests. To analyze categorical variables X2 will be used by Fisher's exact test or Yates correction. A two-tailed test with a p value < 0.05 will be considered as statistically significant. Logistic regression analysis will be used to select independent predictors in those variables that by univariate regression analysis had obtained a p value < 0.01. To avoid confusion, the relationship between historical variables for atherosclerosis and cardiovascular events will be examined through logistic regression and multivariate analysis. Cox proportional risk multivariate model will assess the relationship between each of these variables. Kaplan-Meier survival curves and Cox proportional risk model will be used for adjust survival analysis. A p value < 0.05 will be considered as statistically significant. Data will be expressed as percentages, mean, standard deviation, odds ratio and CI.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 2 years with: a) diagnosis of PH (PAH by RHC), b) Groups I and IV

Exclusion Criteria:

* Severe pulmonary function abnormalities (vital capacity < 60% predicted, FEV1 < 50% predicted)
* Abnormal pulmonary capillary wedge pressure (> 15 mmHg)
* Refusal to participate.

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mexican patients older than 2 years with diagnosis of Pulmonary Hypertension from groups I and IV
Sampling Method: Probability Sample
Enrollment: 875 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 4 years
  In-hospital or outpatient heart failure, cardiogenic shock, syncope, cardiovascular death and bleeding complications.

SECONDARY OUTCOMES:
Cardiovascular death | 4 years
  Secondary to right heart failure, cardiogenic shock, auricular or ventricular arrhythmia.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Sandoval, MD, Principal Investigator — Instituto Nacional de Cardiologia